CLINICAL TRIAL: NCT05223907
Title: Safety and Efficacy of Maintenance of Etomidate Combined With Sevoflurane in General Anesthesia: a Multi-center Randomized Controlled Study
Brief Title: Safety and Efficacy of Maintenance of Etomidate in General Anesthesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ytmz
Record Dates: First submitted 2021-12-28; First posted 2022-02-04 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: General Anesthesia
Keywords: etomidate; propofol; anesthesia maintenance; sevoflurane; anesthesia quality
MeSH Terms: interventions — Etomidate; Propofol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Etomidate (Experimental): Etomidate will be used for general anesthesia
  Interventions: Drug: Etomidate
- Group Propofol (Experimental): Propofol will be used for general anesthesia
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Etomidate — Etomidate will be used for general anesthesia
  Other Names: Etomidate Injectable Emulsion; Yituomizhi, H20020511, WS-400(X-338)-2002-2015Z,YT211101
  Arms: Group Etomidate
Drug: Propofol — Propofol will be used for general anesthesia
  Other Names: Diprivan, JX20060102，H20080473，RW981
  Arms: Group Propofol

SUMMARY:
This study was designed to use etomidate combined with sevoflurane intravenously to maintain anesthesia process under the monitoring of BIS. Propofol was used as the controls. Blood pressure and heart rate were recorded during operation. The VAS pain score was observed after surgery.To investigate whether this program can better maintain intraoperative hemodynamic stability, improve the quality of recovery, and reduce the incidence of postoperative adverse reactions.

ELIGIBILITY:
Inclusion Criteria:

* 18 ≤age≤65;
* Types of surgery: laparoscopic gynecological surgery, laparoscopic gastrointestinal surgery, thoracoscopic radical lung cancer surgery;
* 1 h ≤ operation time ≤ 3 h;
* ASA grade I~III;
* BMI of 18.5~29.9 kg/m2 [BMI= weight (kg)/height (m) 2] (2013 American guidelines for the Management of Overweight and Obesity in Adults);
* In accordance with ethics, the patient voluntarily took the test and signed the informed consent.

Exclusion Criteria:

* Cerebral vascular accident, such as stroke, transient ischemic attack (TIA), etc. within 3 months;
* Severe abnormal liver and kidney function (severe abnormal liver function: ALT, AST, ALP, total bilirubin, one of which is more than 2 times the upper limit of normal value. Severe renal dysfunction: creatinine > 2 times upper normal);
* Patients with diabetic complications (diabetic ketoacidosis, hyperotonic coma, various infections, macrovascular disease, diabetic nephropathy, retinopathy, diabetic cardiomyopathy, diabetic neuropathy, diabetic foot, etc.);
* Unstable angina pectoris or myocardial infarction occurred within 3 months;
* Preoperative blood pressure ≥160/100 mmHg ( ≥ Grade 2 hypertension, 2020 ISH Hypertension Guidelines);
* Identified/suspected abuse or long-term use of narcotic sedatives and analgesics; •Taking hormones or other immunosuppressive agents for more than 10 days within half a year, or having a history of adrenocortical suppression or immune system diseases;
* Hypothyroidism;
* Patients with a history of asthma;
* Those who were reoperated within 3 months;
* Having contraindications or allergies to test drugs and other narcotic drugs;
* Patients enrolled in other studies within 30 days.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1080 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Rate of intraoperative hypertension and hypotension | From the beginning to the end of surgery
  Investigators will record the rate of hypertension and hypotension of participants during intraoperative period
Ricker sedation-agitation score after surgery | 1 day (The period during patients wake up after surgery and general anesthesia in the recovery room.)
  Investigators will record the Ricker sedation-agitation score of participants during recovery period after general anestesia

SECONDARY OUTCOMES:
Postoperative pain scores measured by VAS score. | One-three days after surgery.
  Postoperative pain scores of participants will be assessed by using VAS score (0= no pain, 10= worse pain imaginable)
The incidence of PONV | One-three days after surgery.
  The incidence of postoperative nausea and vomiting of participants will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Zhang, PHD, Study Chair — Henan Provincial People's Hospital
Locations (1):
- Henan Provincial People's Hospital, Zhengzhou, Henan, China